CLINICAL TRIAL: NCT05486546
Title: Comparison of Visual Acuity and Quality of Life Following Contoura With Phorcides Compared to WaveLight Wavefront Optimized LASIK
Brief Title: Contoura With Phorcides Compared to Wavefront Optimized LASIK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Terveen (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor-Investigator, Daniel Terveen, Principal Investigator, Vance Thompson Vision
Organization: Vance Thompson Vision (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMPLIO
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Myopia; Astigmatism
Keywords: Visual acuity; Refractive outcome; LASIK; Contrast sensitivity; Wavefront Optimized; Topography-guided
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study: Phorcides (Experimental): Contoura with Phorcides used for surgical planning of LASIK procedure
  Interventions: Procedure: Contoura with Phorcides
- Control: Wavefront Optimized (Active Comparator): WaveLight Wavefront Optimized used for surgical planning of LASIK procedure
  Interventions: Device: WaveLight Wavefront Optimized

INTERVENTIONS:
Procedure: Contoura with Phorcides — Participants that undergo LASIK surgery using Contoura with Phorcides Analytic Engine
  Arms: Study: Phorcides
Device: WaveLight Wavefront Optimized — Participants that undergo LASIK surgery using WaveLight Wavefront Optimized
  Arms: Control: Wavefront Optimized

SUMMARY:
Comparing post-operative visual acuity and patient reported satisfaction between Contoura with Phorcides and WaveLight Wavefront Optimized.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least age 21 years of age undergoing LASIK eye surgery
* Willing and able to comprehend informed consent and complete 1 month post-op visit
* Potential postoperative BCDVA of 20/20 or better in each eye based on Investigator's medical opinion
* Candidates for Contoura with Phorcides (Myopic, astigmatism <3.0D)
* Both eyes targeted for plano
* Pre-operative total corneal Pachymetry 490um or above
* Stable refractive error <0.50D change in preceding year
* Good general and ocular health
* Pre-operative exam completed within three months of surgery
* SCL discontinued 3 days prior to pre-op exam and the procedure
* Pachymetry above 490 with residual greater than 270um
* Candidates who, as determined by the investigator, can safely undergo LASIK

Exclusion Criteria:

* Patients under 21 years of age
* Concomitant ocular condition which would limit the BCVA at the discretion of the surgeon
* Patients with usual relative and absolute contraindications for LASIK surgery (Patients with severe dry eye, recurrent corneal erosion, uncontrolled Glaucoma, collagen vascular disorders, keratoconus or signs of keratoconus, uncontrolled Diabetes, Herpes)
* Pachymetry below 490
* Autoimmune or immunodeficiency diseases
* Pregnant or nursing women
* Patients with signs of inability to understand consent for study and procedure planned
* Patients with history of previous ocular surgery
* Patients with strabismus or amblyopia
* Patients that have a BCDVA of 20/25 or worse in either eye

Ages: 21 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Post-Op UDVA | 3 months post-op
  Percent of participants with monocular UDVA of 20/16 or better

SECONDARY OUTCOMES:
Post-OP BCVA | 3 months post-op
  Percent of participants with monocular and binocular BCVA of 20/16 or better
Residual Refractive Error | 3 months post-op
  Residual astigmatism and residual SE
Low Contrast Visual Acuity | 3 months post-op
  25% low contrast visual acuity post-op
Pre-op and post-op visual acuity | 3 months post-op
  Percent of participants with post-op UDVA equal to or better than their pre-op CDVA
Corrected Distance Visual Acuity | 3 months post-op
  Compare percent of participants with post-operative and pre-operative CDVA

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Vance Thompson Vison, Bozeman, Montana
  - Vance Thompson Vision, Omaha, Nebraska
  - Vance Thompson Vision, Fargo, North Dakota
  - Vance Thompson Vision, Sioux Falls, South Dakota